CLINICAL TRIAL: NCT03626324
Title: Clinical Evaluation of Connected Catheter 2P (C2P) Wireless Urinary Prosthesis for Management of Neurogenic Lower Urinary Tract Dysfunction
Brief Title: Connected Catheter (C2P) Study for Bladder Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spinal Singularity (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: C2P-01
Record Dates: First submitted 2018-07-26; First posted 2018-08-13 (Actual); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: Urinary Retention; Neurogenic Bladder
Keywords: Spinal Cord Injury (SCI); Neurogenic Lower Urinary Tract Dysfunction (NLUTD); Catheter associated Urinary Tract Infection (CAUTI); Urinary Catheters; Dementia; Stroke; Diabetes; Parkinson's
MeSH Terms: conditions — Urinary Retention; Urinary Bladder, Neurogenic; Spinal Cord Injuries; Dementia; Stroke; Diabetes Mellitus; Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- C2P Study (Experimental): Clinical Evaluation of Connected Catheter 2P Urinary Prosthesis for Management of Neurogenic Lower Urinary Tract Dysfunction
  Interventions: Device: C2P

INTERVENTIONS:
Device: C2P — The C2P is a fully internal, urethral indwelling urinary prosthesis designed for improved bladder management in males with urinary retention disorders requiring catheterization, including neurogenic lower urinary tract dysfunction (NLUTD - e.g. due to spinal cord injury). The C2P is a sterile, single-extended-use device that resides fully internally to the male lower urinary tract (urethra + bladder neck) for an intended service life of up to 29 days per Catheter.

SUMMARY:
The objective of this study is to evaluate the safety and essential performance of the C2P System in males with neurogenic lower urinary tract dysfunction (NLUTD), both in an acute clinical setting and an extended period of home use.

DETAILED DESCRIPTION:
Spinal Singularity had developed C2P system to address several drawbacks of current standard-of-care urinary catheters. The C2P is fully internal, urethral indwelling urinary prosthesis designed for improved bladder management in males with urinary retention disorders requiring catheterization, including NLUTD. The C2P is a sterile, single-extended use device that resides fully internally to the male lower urinary tract for an intended service life of up to 29 days per catheter

ELIGIBILITY:
Inclusion Criteria:

1. Males age ≥ 18 with clinical diagnosis of neurogenic lower urinary tract dysfunction (NLUTD)
2. Must be clinically suitable and capable of safely managing bladder using an intermittent voiding or indwelling strategy

   * Must have stable urinary management history: no significant changes in bladder management regimen within past 12 months

   OR:
   * Must have urodynamic profile suitable for C2P, as assessed via urodynamics study within past 12 months (including bladder capacity > 200mL without uninhibited bladder contractions)
3. Subject's lower urinary tract anatomy must fall within the ranges serviceable by the C2P device, as specified in the investigational device instructions for use (IFU).

Exclusion Criteria:

1. Active symptomatic urinary tract infection, as defined in this protocol (subjects may receive the device after Urinary Tract Infection (UTI) has been treated)
2. Significant risk profile or recent history of urethral stricture (e.g. stricture within past 90 days)
3. Significant risk profile or recent history of clinically significant autonomic dysreflexia (AD) (e.g. History of hospitalization due to AD within past 12 months)
4. Significant intermittent urinary incontinence (between catheterizations)
5. Uninhibited bladder contractions and/or vesico-ureteral reflux that is not reliably controlled with medication or alternate therapy (e.g. Botox injections)
6. Pre-existing urinary pathologies and/or morphological abnormalities of the lower urinary tract or bladder (assessed during in-depth medical screening, including cystoscopy and urine analysis)
7. Urinary tract inflammation or neoplasm
8. Urinary fistula
9. Bladder diverticulum (outpouching) > 5cm in size
10. Chronic pyelonephritis (secondary to upper urinary tract infection(s) within past 6 months)
11. Impaired kidney function or renal failure
12. Active gross hematuria
13. Active urethritis
14. Bladder stones
15. Dependence on an electro-magnetic medical implant (e.g. cardiac pacemaker or implanted drug pump) or external device
16. Any unsuitable comorbidities as determined by the investigator or complications related to use of certain medications
17. Any physical or cognitive impairments that diminish the subject's ability to follow directions or otherwise safely use the C2P System

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 27 (Actual)
Dates: Start 2018-07-25 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Freedom from genito-urinary injury/trauma | 3 months
  Improved bladder management without injury to genito-urinary tract
Successful Acute Performance- I | Day 0 (On the day of C2P insertion)
  To evaluate successful retention of C2P
Successful Acute Performance- II | Day 0 (On the day of C2P insertion)
  To evaluate successful bladder voiding with C2P
Successful Acute Performance- III | Day 0 (On the day of C2P insertion)
  To evaluate successful valve sealing of C2P
Successful Home-use Performance | 3 months
  To evaluate successful home use of C2P using same measures as Acute Performance

CONTACTS AND LOCATIONS:
Overall Officials: Derek Herrera, Study Director — Spinal Singularity
Locations (8):
- United States (8):
  - Northwest Urology Associates, 9151 West Thunderbird Rd, Suite 104, Peoria, Arizona
  - Northwest Urology Associates, 14674 W. Mountain View Blvd, Suite 210, Surprise, Arizona
  - West Coast Urology, 11411 Brookshire Avenue, Suite 508, Downey, California
  - West Coast Urology, 575 E. Hardy St., Suite 215, Inglewood, California
  - Tri Valley Urology, 25495 Medical Center Dr., Suite 204, Murrieta, California
  - Minnesota Urology, 6025 Lake Road Suite 200, Woodbury, Minnesota
  - New Jersey Urology, 15000 Midlantic Drive, Suite 100, Mount Laurel, New Jersey
  - New Jersey Urology, 2401 Evesham Road, Suite F, Voorhees Township, New Jersey